CLINICAL TRIAL: NCT04828473
Title: Green Light Effect on Sleep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Green Light Study Center (Other)
Responsible Party: Principal Investigator, Paul Hart, Primary Care Provider, The Green Light Study Center
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 001
Record Dates: First submitted 2021-03-27; First posted 2021-04-02 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: single group assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Allay Lamp — The Allay Lamp is a consumer product currently available and widely used in the US. It emits low intensity (1-10lux)narrow band (20nm) green light (peak wavelength 520nm) that is marketed as non-irritating to users. In that context, it is not a medical device and does not require a 510(k). However, we believe that light likely also has benefits for sleep. To better understand its effects,we are planning to conduct the proposed study. In that context, the Allay Lamp would be considered an investigational medical device because it has not been cleared or approved by FDA for the intended purpose of treating sleep. No FDA submission should be necessary for this study using 21 C.F.R. 812.3, because the Allay Lamp is a non-significant risk (NSR) device:
  * It is not an implant
  * It is not intended for use in supporting or sustaining human life The Allay Lamp provides a very low risk light-based therapy. The light provides no more risk than any other table lamp available on the market today.

SUMMARY:
The main goal of this study is to determine whether exposure to a narrow band of green light (NBGL) improved sleep quality in healthy subjects.

This is a within-subject study design that examines NBGL effects on sleep onset, sleep fractures (i.e., how many times per night the subjects wake up), total sleep duration, and sleep quality using high-resolution assessments. To complete the study, each participant will complete a 30-day, daily sleep diary while using white light (i.e., being in regular room light) during the last 2 hours of their waking period. This period will be defined as the baseline/control arm of the study. After completing this phase 1, subjects will receive a lamp designed to emit the narrow band of green light and again be asked to complete a 30-day, daily sleep diary, but this timer while using the NBGL light (i.e., being in what appears green light) during the last 2 hours of their waking period. This period will be defined as the active arm of the study. After completing this phase 2,

DETAILED DESCRIPTION:
Sleep quality will be assessed using the Consensus sleep diary [Carney et al., (2012)] The consensus sleep diary: Standardizing prospective sleep self-monitoring, Sleep Vol.35, No.2, pp.287-302], the latter of which captures total sleep time, sleep latency, wake after sleep onset, number of awakenings, quality, sleep efficiency, and trouble staying awake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who wish to improve their sleep quality

Exclusion Criteria:

* Subjects diagnosed with sleep disorders and are currently on medications and/or devices that aid their sleep ( eg trazadone as medication, CPAP)

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
narrow band green light and sleep | 2 months
  this primary outcome measures improvement in sleep quality during the month in which subjects used the green light as compared to the month in which they used the regular room light. Sleep quality will be measured by the Consensus Sleep Diary. THe Consensus Sleep Diary requires subjects to answer 8 questions by depicting numbers that represent best their answers. These numbers provide the basis for our ability to quantify the difference between the two light conditions of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Green Light Sleep Study Center, Boca Raton, Florida, United States